CLINICAL TRIAL: NCT06723691
Title: A Single Center, Open-label, Two Cohorts, Fixed Sequence Trial, Investigating the Influence of HRS9531 Injection on Gastric Emptying and Pharmacokinetics of Metformin, Atorvastatin, Warfarin, and Digoxin in Healthy Subjects
Brief Title: Influence of HRS9531 on Gastric Emptying and Pharmacokinetics of Metformin, Atorvastatin, Warfarin, and Digoxin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS9531-107
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acetaminophen; Metformin; Warfarin; Atorvastatin; Digoxin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Drug: Acetaminophen; Drug: Metformin; Drug: Warfarin; Drug: Atorvastatin; Drug: Digoxin; Drug: HRS9531

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen
Drug: Metformin — Metformin
Drug: Warfarin — Warfarin
Drug: Atorvastatin — Atorvastatin
Drug: Digoxin — Digoxin
Drug: HRS9531 — HRS9531

SUMMARY:
The purpose of this study is to evaluate the influence of HRS9531 injection on gastric emptying and pharmacokinetics of metformin, atorvastatin, warfarin, and digoxin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, be able and willing to provide a written informed consent;
2. Male subjects aged 18-45 years on the date of signing informed consent (inclusive);
3. Body weight ≥60 kg, body mass index (BMI) within the range of 24.0-35.0 kg/m2 (inclusive);
4. HbA1c<6.0%;
5. The subjects have no plans to have children and voluntarily take effective contraceptive measures from the time of signing the informed consent to 2 months after the last medication, and have no plans to donate eggs/sperm; the pregnancy test of female subjects with fertility must be negative.

Exclusion Criteria:

1. Chronic or severe medical history of the respiratory system, circulatory system, digestive system, urinary system, blood system, endocrine system, immune system, nervous system, mental system, etc., or those with existing systemic diseases mentioned above, and judged by the investigator to be unsuitable to participate in this study;
2. Past history or family history of medullary thyroid cancer or multiple endocrine neoplasia type 2 (MEN2), a history of pancreatitis or symptomatic gallbladder stones;
3. History of disease that increases the risk of bleeding;
4. Surgery within 6 months prior to dosing, planned to undergo surgery during the study period;
5. Participation in clinical trials of any drug or medical device in the 3 months or 5 half-lives, whichever longer, prior to dosing;
6. Blood donation history or blood loss ≥400 mL within 3 months or ≥200 mL within 1 month before dosing, or received blood transfusion within 3 months before dosing;
7. Hepatitis B surface antigen (HBsAg), HIV antibody, hepatitis C virus antibody (HCVAb), treponema pallidum specific antibody detection, positive;
8. Abnormal laboratory test results or abnormal examinations considered unsuitable to participate in this trial;
9. History of hypoglycaemia;
10. History of syncope or vasovagal episodes, difficulty with blood collection, or an inability to tolerate venipuncture;
11. The investigator considers that the subject has any other factors that would make it inappropriate to participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2025-06-09 (Actual)

PRIMARY OUTCOMES:
Area under the acetaminophen plasma concentration-time curve | From time 0 to 24 hours after a single dose.
Maximum observed acetaminophen concentration | From time 0 to 24 hours after a single dose.
Time of maximum observed acetaminophen concentration | From time 0 to 24 hours after a single dose.
Area under the metformin plasma concentration-time curve | From time 0 to 12 hours after the last of 7 repeated doses.
Area under the S-warfarin plasma concentration-time curve | From time 0 to 168 hours after a single dose.
Area under the atorvastatin plasma concentration-time curve | From time 0 to 72 hours after a single dose.
Area under the digoxin plasma concentration-time curve | From time 0 to 120 hours after a single dose.

SECONDARY OUTCOMES:
Area under the concentration versus time curve of acetaminophen from 0 to infinity | Start of treatment up to 168 hours.
Apparent volume of distribution of acetaminophen | Start of treatment up to 168 hours.
Time of maximum observed metformin concentration after 3.5 days of treatment | Start of Treatment up to 30 hours.
Clearance of metformin after 3.5 days of treatment | Start of Treatment up to 30 hours.
Apparent volume of distribution of metformin after 3.5 days of treatment | Start of Treatment up to 30 hours.
Time of maximum observed S-warfarin concentration | Start of Treatment up to 168 hours.
Clearance of S-warfarin | Start of Treatment up to 168 hours.
Apparent volume of distribution of S-warfarin | Start of Treatment up to 168 hours.
Time of maximum observed atorvastatin (and its active metabolites) concentration | Start of Treatment up to 72 hours.
Clearance of atorvastatin (and its active metabolites) | Start of Treatment up to 72 hours.
Time of maximum observed digoxin concentration | Start of Treatment up to 120 hours.
Maximum observed digoxin concentration | Start of Treatment up to 120 hours.
Clearance of digoxin | Start of Treatment up to 120 hours.
Apparent volume of distribution of digoxin | Start of Treatment up to 120 hours.
Time of maximum observed HRS9532 concentration | Start of Treatment up to 168 hours.
Maximum observed HRS9531 concentration | Start of Treatment up to 168 hours.
Area under the concentration versus time curve of HRS9531 from 0 to the time of the last measurable (positive) concentration | Start of Treatment up to 168 hours.
Area under the concentration versus time curve of HRS9531 from 0 to infinity | Start of Treatment up to 168 hours.
Incidence and severity of adverse events | Screening period up to 117 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided